CLINICAL TRIAL: NCT07069920
Title: Single-center, Randomized, Subject/Evaluator-blinded, Split-face, Active-controlled, Non-inferiority, Pivotal Clinical Trial to Compare the Safety and Efficacy Between BRDE33-100 and the Soonsoofill in Temporary Correction of Moderate to Severe Nasolabial Folds
Brief Title: To Evaluate the Efficacy and Safety of 'BRDE33-100' for the Temporary Correction of Moderate to Severe Nasolabial Folds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BRPharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Revitrane HA24-01
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Nasolabial Folds
Keywords: Nasolabial folds; Hyaluronic acid filler; Dermal Filler; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The experimental group (Experimental): BRDE33-100
  Interventions: Device: BRDE33-100
- The control group (Active Comparator): Soonsoofill
  Interventions: Device: Soonsoofill

INTERVENTIONS:
Device: BRDE33-100 — BRDE33-100 will be injected once at Visit 2 (Baseline).
  Arms: The experimental group
Device: Soonsoofill — Soonsoofill will be injected once at Visit 2 (Baseline).
  Arms: The control group

SUMMARY:
This study aims to demonstrate the non-inferiority of BRDE33-100 to Soonsoofill in temporarily improving moderate to severe nasolabial folds.

DETAILED DESCRIPTION:
This confirmatory clinical trial aims to demonstrate the non-inferiority of 'BRDE33-100' by comparing and evaluating the efficacy and safety of 'BRDE33-100' with 'Soonsoofill'.

This study follows a split-face design in which both the investigational device and the control device are used for treatment in each subject-one on each nasolabial fold. Device allocation will be determined by opening sealed randomization envelopes prior to each treatment. Efficacy and safety assessments will be conducted for 24 weeks after the initial treatment, followed by an additional 24-week long-term follow-up period, for a total participation duration of 52 weeks. Efficacy assessments will include the Wrinkle Severity Rating Scale (WSRS), the Global Aesthetic Improvement Scale (GAIS), and a pain evaluation using the Visual Analogue Scale (VAS). Safety assessments will include adverse event monitoring, clinical laboratory testing, vital signs, and physical examinations. At each efficacy assessment visit, including the baseline, standardized photographs of the treatment area will be taken, and WSRS scoring will be performed by an independent evaluator based on these images.

ELIGIBILITY:
Inclusion Criteria: All of the following inclusion criteria must be met for a subject to be enrolled in this clinical trial.

* Male or female subjects aged between 19 and 75 years, inclusive, as of the date of written informed consent.
* Voluntarily decided to participate in the study and signed the informed consent form in writing
* Subjects who desire improvement in nasolabial folds and have a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4.
* Subjects whose bilateral nasolabial folds appear visually symmetrical, although WSRS scores do not need to be identical on both sides.
* Subjects who agree to use appropriate contraception from the date of signing the informed consent form until 3 months after the end of the clinical trial. *Examples of acceptable contraception include: copper intrauterine device (IUD), hormone-releasing IUD, condoms, vasectomy, tubal ligation, spermicides, vaginal contraceptive film, subdermal implants, injectable contraceptives, female condoms, and oral contraceptives.
* Subjects who agree not to undergo any procedures or treatments that may affect the nasolabial folds during the study period.
* Subjects who are able to understand and comply with the study instructions and are available for the entire duration of the study.

Exclusion Criteria: Subjects who meet any of the following exclusion criteria will not be eligible for participation in this clinical trial.

* Received antithrombotic agents (except for low-dose aspirin [100 mg, up to 300 mg/day]) or nonsteroidal anti-inflammatory drugs (NSAIDs) within 2 weeks prior to screening
* Used topical agents on the device application area within 4 weeks prior to screening or plans to use them during the study period, including corticosteroids, retinoids, alpha hydroxy acids, skin-whitening agents, or anti-wrinkle functional cosmetics. (- Topical corticosteroids for therapeutic purposes may be used for a short duration of up to 14 consecutive days.)
* Received invasive laser treatment, deep peeling procedures, or filler injections on the device application area within 24 weeks prior to screening.
* Received any wrinkle improvement procedures on the device application area within 24 weeks prior to screening, including:

  * Botulinum toxin injections
  * Soft-tissue augmentation
  * Facial lifting surgery
  * Dermabrasion
  * Dermal photo-rejuvenation
* Received any wrinkle improvement procedures on the device application area within 1 year prior to screening, including facial augmentation using calcium hydroxylapatite or wrinkle treatment using approved fillers.
* Received an injection of calcium hydroxylapatite in the nasolabial fold area within 1 year prior to screening.
* Has permanent dermal implants such as Softform or silicone in the nasolabial fold area.
* Underwent facial lifting involving thread-based tissue fixation (e.g., thread lifting) that affected the nasolabial fold area within 1 year prior to screening
* Has taken medications that may affect skin hypersensitivity testing, including:

  ① First- or second-generation antihistamines (e.g., chlorpheniramine, hydroxyzine, cetirizine, fexofenadine, loratadine) within 7 days prior to screening

  ② Tricyclic antidepressants (e.g., imipramine, doxepin) within 11 days prior to screening

  ③ H2-receptor antagonists (e.g., ranitidine) within 1 day prior to screening
* Has scars, skin disorders, wounds, infections, inflammation, or other skin lesions in the nasolabial fold area that may affect the outcome of this clinical trial.
* Has a history of anaphylaxis or severe systemic allergic reactions.
* Has a history of hypertrophic scarring, keloid formation, or hyperpigmentation.
* Has a known hypersensitivity to Hyaluronic acid (HA).
* Has experienced adverse reactions to EMLA Cream or other lidocaine-based anesthetic products.
* Has or has had autoimmune diseases including AIDS, or is immunocompromised.
* Has clinically significant disorders of the cardiovascular, gastrointestinal, respiratory, endocrine, or central nervous systems, or has psychiatric conditions that may affect participation in this clinical trial.
* Tested positive on the skin hypersensitivity test indicating hypersensitivity to the investigational device or control device at the time of screening.
* Participated in other clinical trial(s) within 30 days prior to screening
* Pregnant or breast-feeding women (women of childbearing potential must undergo a pregnancy test)
* Subjects who, due to physical, neurological, or psychological conditions, are unable to comply with all aspects of the screening, evaluation, treatment, and follow-up schedule.
* Subjects who are otherwise unable to communicate or follow instructions properly.
* Determined by the principal investigator to be unable to participate in the study for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Wrinkle Severity Rating Scale (WSRS) score from baseline to Week 24 after the final treatment with the investigational device, as assessed by an independent evaluator | Baseline, Week 24
  The Wrinkle Severity Rating Scale (WSRS) is a five-point grading scale ranging from 5 (extreme deep nasolabial folds) to 1 (no visible nasolabial folds). An independent evaluator assesses wrinkle severity based on photographs of the treatment area, while the investigator performs a direct visual evaluation of the same site. For the independent assessment, photographs of the nasolabial folds taken under normal lighting from the front, left, and right angles are used for evaluation.

SECONDARY OUTCOMES:
Change in WSRS score from baseline to Weeks 8, 16, 36, and 48 after the treatment with the investigational device, as assessed by an independent evaluator | Baseline, Weeks 8, Weeks 16, Weeks 36, Weeks 48
  The Wrinkle Severity Rating Scale (WSRS) is a five-point grading scale ranging from 5 (extreme deep nasolabial folds) to 1 (no visible nasolabial folds). An independent evaluator assesses wrinkle severity based on photographs of the treatment area, while the investigator performs a direct visual evaluation of the same site. For the independent assessment, photographs of the nasolabial folds taken under normal lighting from the front, left, and right angles are used for evaluation.
Change in WSRS score from baseline to Weeks 8, 16, 36, and 48 after the final treatment with the investigational device, as assessed by the investigator | Baseline, Weeks 8, Weeks 16, Weeks 36, Weeks 48
  The Wrinkle Severity Rating Scale (WSRS) is a five-point grading scale ranging from 5 (extreme deep nasolabial folds) to 1 (no visible nasolabial folds). An independent evaluator assesses wrinkle severity based on photographs of the treatment area, while the investigator performs a direct visual evaluation of the same site. For the independent assessment, photographs of the nasolabial folds taken under normal lighting from the front, left, and right angles are used for evaluation.
Global Aesthetic Improvement Scale (GAIS) score assessed by the investigator at Weeks 8, 16, 36, and 48 after the final treatment | Weeks 8, Weeks 16, Weeks 36, Weeks 48
  The Global Aesthetic Improvement Scale (GAIS) is a post-treatment assessment scale ranging from 3 (very much improved) to -1 (worse). It is used to evaluate the degree of aesthetic improvement by directly observing the treated area at each time point in comparison to the pre-treatment condition.
Global Aesthetic Improvement Scale (GAIS) score assessed by the subject at Weeks 8, 16, 36, and 48 after the final treatment | Weeks 8, Weeks 16, Weeks 36, Weeks 48
  The Global Aesthetic Improvement Scale (GAIS) is a post-treatment assessment scale ranging from 3 (very much improved) to -1 (worse). It is used to evaluate the degree of aesthetic improvement by directly observing the treated area at each time point in comparison to the pre-treatment condition.
Proportion of subjects showing a reduction of ≥1 point in WSRS score from baseline, as assessed by an independent evaluator at Weeks 8, 16, 36, and 48 after the final treatment | Baseline, Weeks 8, Weeks 16, Weeks 36, Weeks 48
  The Wrinkle Severity Rating Scale (WSRS) is a five-point grading scale ranging from 5 (extreme deep nasolabial folds) to 1 (no visible nasolabial folds). An independent evaluator assesses wrinkle severity based on photographs of the treatment area, while the investigator performs a direct visual evaluation of the same site. For the independent assessment, photographs of the nasolabial folds taken under normal lighting from the front, left, and right angles are used for evaluation.
Proportion of subjects showing a reduction of ≥1 point in WSRS score from baseline, as assessed by the investigator at Weeks 8, 16, 36, and 48 after the final treatment | Baseline, Weeks 8, Weeks 16, Weeks 36, Weeks 48
  The Wrinkle Severity Rating Scale (WSRS) is a five-point grading scale ranging from 5 (extreme deep nasolabial folds) to 1 (no visible nasolabial folds). An independent evaluator assesses wrinkle severity based on photographs of the treatment area, while the investigator performs a direct visual evaluation of the same site. For the independent assessment, photographs of the nasolabial folds taken under normal lighting from the front, left, and right angles are used for evaluation.
Mean pain score assessed by the subject using a 100 mm visual analogue scale (VAS) at 30 minutes after the initial treatment with the investigational device | Baseline
  The Visual Analog Scale (VAS) is a 100 mm vertical line with the left end labeled as "no pain (0 points)" and the right end labeled as "unbearable pain (10 points)." The subject marks a point on the line to indicate their perceived level of pain, and the distance from the 0-point to the marked line is measured in millimeters. The score is recorded in 1 mm increments, with lower scores indicating less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jiye Kim, M.D., PhD, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Name: Wonju severance Christian hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No